CLINICAL TRIAL: NCT05638152
Title: Effect of a Bundle of Non-pharmacological Interventions on the Stress Response to Surgery
Acronym: SPACU-lab
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N22SCL
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-11

CONDITIONS: Surgical Injury; Stress, Physiological; Stress, Psychological; Pain, Postoperative
Keywords: non-pharamacological; analgesia; stress; postoperative; surgical stress response; post anesthesia care unit
MeSH Terms: conditions — Intraoperative Complications; Stress, Psychological; Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (3x 15 ml) for cortisol, IL-6, CRP, glucose, neutrophil-lymphocyte ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before: routine care
- after: routine care + natural imagery in the PACU + access to music + access to aromatherapy + use of hypnoidal communication techniques by PACU nurses
  Interventions: Other: implementation of a bundle of non-pharmacological interventions aimed at stress reduction

INTERVENTIONS:
Other: implementation of a bundle of non-pharmacological interventions aimed at stress reduction — The bundle consists of 4 interventions:
  * natural imagery in the PACU (wall length decorations and lighted ceiling panels with sky views
  * Aromatherapy with fragrances selected for anxiolytic and antiemetic properties
  * Music available to patients
  * Comfort Talk communication course for PACU nurses
  Groups: after

SUMMARY:
Rationale: Surgical trauma and post-surgical pain induce a physiological stress response that can be detrimental to the patient. Non-pharmacological interventions aimed at stress reduction are known to reduce pain scores and opioid consumption. The effect of these interventions on the surgical stress response are unknown.

Objective: To assess the effect of a bundle of non-pharmacological interventions implemented in the post-anesthesia care unit on the total serum cortisol levels after intermediate and major surgery.

Study design: This is a prospective before-after study. Study population: Patients scheduled for intermediate or major oncological surgery in a tertiary referral cancer center.

Intervention: The implementation of a bundle of four non-pharmacological interventions aimed at stress reduction in the post-anesthesia care unit. The bundle consists of: access to music, aromatherapy, natural images on the walls and ceiling and communication techniques aimed at reduction of stress and pain.

Main study parameters/endpoints: Serum cortisol levels on the first postoperative day.

DETAILED DESCRIPTION:
This protocol is a substudy of a larger observational before-after study that studies the effects of the planned implementation of a bundle of non-pharmacological interventions in the post-anesthesia care unit on pain scores, opioid consumption and quality of recovery.

In this current protocol, a subset of 90 surgical patients of a tertiary referral cancer centre in the Netherlands will be included and will be asked to provide informed consent for additional blood samples to be drawn to study the effects of the stress-reducing bundle on biomarkers of the surgical stress response.

45 eligible patients will be approached in the before-arm of the study and 45 will be included for the after-arm. Inclusion criteria are: planned for intermediate to major oncological surgery with an expected duration of >120 minutes, without the use of neuraxial anesthetic techniques. Patients with a planned postoperative ICU-admission will be excluded. After providing informed consent, they will be asked to complete a Quality of Recovery (QoR-15) questionnaire prior to surgery. Additional blood will be drawn with their routine preoperative blood sample on the morning of surgery to determine levels of cortisol, interleukine-6 (IL-6), glucose, C-reactive protein (CRP) and Neutrophil-Lymphocyte Ratio(NLR). The same blood sample will be drawn on arrival in the PACU and on the morning of the first postoperative day. Patients will also be asked to complete the QoR-15 questionnaire again on the first postoperative day.

The primary outcome will be serum cortisol level on the first postoperative day (as a biomarker of the surgical stress response).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* scheduled for intermediate to major oncological surgery
* with a minimum duration of 120 mins

Exclusion Criteria:

* Neuraxial anesthetic technique
* planned for postoperative ICU admission
* day case surgery
* Indication for peri-operative steroids
* chronic use of steroids
* Bronchial hyperreactivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults scheduled for intermediate to major oncological surgery in a tertiary referral cancer centre in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
serum cortisol level on POD1 | 24 hours
  serum cortisol level on postoperative day 1

SECONDARY OUTCOMES:
serum IL-6, glucose, CRP, NLR on POD 1 | 24 hours
  serum IL-6, glucose, CRP, NLR on postoperative day 1

IPD SHARING:
Plan to Share IPD: Undecided